CLINICAL TRIAL: NCT05282160
Title: The Influence of Prepartum Perineal Training With the Epi-No Device on Pelvic Floor Function in Women 6 Months After Delivery.
Brief Title: The Influence of Prepartum Perineal Training With the Epi-No Device on Pelvic Floor Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: ULondrina1
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2020-11

CONDITIONS: Dyspareunia; Urinary Incontinence; Perineal Tear; Perineal Injury; Episiotomy Wound; Episiotomy; Complications
Keywords: Pelvic floor; Epino; Birth; Sexual Function; Continence; Perineum
MeSH Terms: conditions — Dyspareunia; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group (G1) will be composed of puerperal women over 18 years of age attended by Lucila Balalai Municipal Maternity in Londrina. Recruitment will be done through a chart review, which will include single-fetus primiparous that delivered on full term without intercurrence (between 37 and 42 weeks).
- Epino Group (Experimental): The study group (G2) will be composed of women over 18 years of age, primigravidae, between 30 and 32 weeks of gestation attended by the Basic Health Units of the central region of Londrina. Only those who agree to participate in the study and sign the free and informed consent form will be included.
  Interventions: Device: Epino

INTERVENTIONS:
Device: Epino — The pregnant women will perform 10 sessions (twice a week for 5 weeks) of perineal preparation with the Epi-No device (pressure gauge connected to an inflatable soda that simulates the baby's head the vaginal canal). After the introduction of the deflated probe (only the first half of the device), it is minimally inflated until the perception in the vaginal canal. The first 5 minutes will be for perception of the pelvic floor with contraction and relaxation with the purpose of toning and maintaining muscular strength, followed by 15 minutes of perineal elongation respecting the tolerance of the pregnant woman. After 20 minutes in total, the pregnant woman relaxes so that the inflated device leaves gently of her vaginal cavity and the physiotherapist helps at that moment. After the device is removed, note the circumference reached on the day.
  Other Names: perineal preparation
  Arms: Epino Group

SUMMARY:
Perineal injury is the most common maternal obstetric complication associated with vaginal delivery (1). It is estimated that perineal lacerations of first and second degree occur in 38% of spontaneous vaginal deliveries in primiparous and in 36% in multiparous women (2). The perineal traumas are associated with significant maternal morbidity, including pain, urinary and fecal incontinence, genital prolapses, dyspareunia, physical and psychological damage (3,4). Episiotomy is a surgical procedure used in obstetrics to increase vaginal opening with an incision in the perineum at end of the second stage of vaginal delivery. However, this procedure is commonly used improperly as routine in the delivery attendance in many health services. For a successful vaginal delivery, the vaginal opening should slowly dilate in order to allow stretching because when the baby descends rapidly, the tissues can tear (11). The degree of muscle stretching or distension in the vaginal delivery may lead to pelvic floor muscle trauma (12). Urinary incontinence is the involuntary loss of urine, with impacts on women in terms of their quality of life, and is considered a social and hygiene problem (16). The muscle strength of the pelvic floor is important for the prevention, diagnosis and treatment of pelvic floor dysfunction. EPI-NO is a device that was invented by a German obstetrician in order to prepare and train the pelvic floor for normal delivery. The purpose of this study is to verify the effect of 10 sessions of pelvic floor elongation with Epi-No in the prevention of urinary incontinence and dyspareunia 6 months after delivery.

DETAILED DESCRIPTION:
The control group (G1) will be composed of women over 18 years of age attended by Lucila Balalai Municipal Maternity in Londrina. Recruitment will be done through a chart review, which will include single-fetus primiparous that delivered on full term without intercurrence (between 37 and 42 weeks). After birth they will receive project information while still hospitalized and are scheduled for evaluation 5 months after delivery if they consent to participate in the project. The study group (G2) will be composed of women over 18 years of age, primigravidae, between 30 and 32 weeks of gestation attended by the Basic Health Units of the central region of Londrina. Only those who agree to participate in the study and sign the free and informed consent form (Appendix 1) will be included.

Group one will be evaluated before the intervention (between 30th and 32nd week) and 6 months after delivery. The control group will be evaluated only once in the sixth month after delivery. The evaluators will be blind and the evaluation will be composed by:

* Anamnesis containing data on pregnancy and delivery (hours of expulsive period, use of instruments and / or maneuvers, degree of laceration, episiotomy, and characterization of possible urinary or sexual complaints);
* Physical examination: inspection and vaginal palpation in order to verify the capacity of external and internal perineal contraction and tenderness with touch;
* Visual Analogue Scale for dyspareunia included;
* Validated sexual dysfunction assessment questionnaire for Portuguese: Female Sexual Function Index (FSFI) .
* Quality of life questionnaire SF-36.

The pregnant women will perform 10 sessions (twice a week for 5 weeks) of perineal preparation with the Epi-No device (pressure gauge connected to an inflatable soda that simulates the baby's head the vaginal canal). The evaluations and sessions of Epi-No will be individual and will take place in the research laboratory of the physiotherapy outpatient clinic of the University Hospital of Londrina.

The protocol was developed by a group of researchers based on the suggestions of already developed studies and clinical practice. After the introduction of the deflated probe (only the first half of the device), it is minimally inflated until the perception in the vaginal canal. The first 5 minutes will be for perception of the pelvic floor with contraction and relaxation with the purpose of toning and maintaining muscular strength, followed by 15 minutes of perineal elongation respecting the tolerance of the pregnant woman. After 20 minutes in total, the pregnant woman relaxes so that the inflated device leaves gently of her vaginal cavity and the physiotherapist helps at that moment. After the device is removed, note the circumference reached on the day.

After the procedure the pregnant woman sits on the ball and performs some contractions of perineum to relieve the eventual sensation of burning.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women over 18 years of age, attended by the Basic Health Units of the central region of Londrina.

Exclusion Criteria:

* patients with complaint of urinary incontinence or dyspareunia prior to pregnancy, not controled hypertension (SAH) and gestational diabetes, placenta previa, twin pregnancy, who have undergone perineal or vaginal surgeries, who have a urinary tract infection, genital herpes, ongoing candidiasis and any other diagnosis in which the normal delivery becomes a risk.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Urinary Incontinence questionnaire | 6 months after delivery
  score of validated questionnaire
Dyspareunia questionnaire | 6 months after delivery
  score of validated questionnaire

SECONDARY OUTCOMES:
Pelvic floor strength | 6 months after delivery
  number measured by intravaginal perineometry
Quality of life score | 6 months after delivery
  score of validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: SILVIO HM ALMEIDA, DOCTOR, Study Chair — State University of Londrina
Locations (1):
- Universidade Estadual de Londrina, Londrina, Paraná, Brazil